CLINICAL TRIAL: NCT07339397
Title: Incidence and Determinants of Joint Contractures in Mechanically Ventilated Intensive Care Unit Patients: a Prospective Cohort Study
Brief Title: Incidence and Determinants of Joint Contractures in Mechanically Ventilated ICU Patients
Acronym: ICU-CONTRACT
Status: Recruiting | Type: Observational
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Principal Investigator, Oğuz Kağan Bulut, Principal Investigator, Elazıg Fethi Sekin Sehir Hastanesi
Other Study IDs: FSH-ICU-CONTRACTURE-2025
Record Dates: First submitted 2026-01-02; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Joint Contractures; Critical Illness; Mechanical Ventilation; INTANSIVE CARE
Keywords: Joint contracture; Intensive care unit; Mechanical ventilation; Passive range of motion; Musculoskeletal complications; Physiotherapy
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically Ventilated ICU Patients: Adult patients admitted to the intensive care unit who are mechanically ventilated, immobilized, and have impaired consciousness. All participants will receive routine ICU care and standard physiotherapy according to institutional protocols. No additional interventions or experimental procedures will be applied as part of the study.

SUMMARY:
This prospective observational cohort study aims to evaluate the incidence and determinants of joint contracture development in mechanically ventilated adult patients admitted to the intensive care unit (ICU). Prolonged immobilization, deep sedation, and neuromuscular blockade are common in critically ill patients and may contribute to musculoskeletal complications, including joint contractures, which can adversely affect functional outcomes and rehabilitation after ICU discharge.

Adult patients who are mechanically ventilated, immobilized, and have impaired consciousness will be consecutively enrolled and followed during their ICU stay. Joint range of motion will be assessed using standardized passive range of motion (PROM) measurements performed with a goniometer at predefined intervals by trained assessors. Joint contracture will be defined as a reduction of at least 33% in passive joint range of motion compared with normal reference values.

This study is non-interventional, and all patients will receive routine ICU care and standard physiotherapy according to institutional protocols. No additional procedures or interventions will be applied for research purposes. Demographic characteristics, clinical variables, and ICU-related factors will be recorded to explore potential associations with contracture development.

The findings of this study are expected to provide prospective data on the burden of joint contractures in mechanically ventilated ICU patients and to identify modifiable risk factors that may inform future preventive and rehabilitative strategies in critical care practice.

DETAILED DESCRIPTION:
This study is designed as a prospective, non-interventional observational cohort study conducted in a tertiary-level intensive care unit (ICU). The primary objective is to determine the incidence of newly developed joint contractures and to identify clinical and ICU-related factors associated with contracture development in mechanically ventilated adult patients.

Adult patients (≥18 years) who are mechanically ventilated, immobilized, and have impaired consciousness will be consecutively enrolled within the first 48 hours of ICU admission. Patients will be followed throughout their ICU stay. Individuals with pre-existing joint contractures, amputations, neuromuscular diseases, spasticity, or conditions preventing safe joint assessment will be excluded.

Joint range of motion will be evaluated using standardized passive range of motion (PROM) measurements performed with a goniometer. Measurements will be conducted at predefined intervals, twice weekly, by trained physiotherapists or physical medicine specialists. The same evaluator and consistent time windows will be used whenever possible to ensure measurement reliability. Joint contracture will be defined as a reduction of at least 33% in passive joint range of motion compared with established normal reference values.

All patients will receive routine ICU care, including standard physiotherapy practices such as positioning, passive or active-assisted joint exercises, respiratory physiotherapy, and early mobilization when clinically appropriate. No additional interventions, treatments, or procedures will be introduced for research purposes.

Demographic data, clinical characteristics, and ICU-related variables-including duration of mechanical ventilation, length of ICU stay, sedation duration, use of neuromuscular blocking agents, timing of mobilization, severity scores, and clinical outcomes-will be prospectively recorded.

Descriptive statistics will be used to summarize patient characteristics and contracture incidence. Comparative analyses will be performed between patients with and without joint contracture development. Multivariable regression models will be used to explore independent factors associated with contracture development. Time-to-event analyses may be applied to evaluate the timing of contracture occurrence during the ICU stay.

The results of this study are expected to provide robust prospective data on the burden and determinants of joint contractures in mechanically ventilated ICU patients, thereby contributing to improved preventive and rehabilitative strategies in critical care.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients aged 18 and over

  * Patients on mechanical ventilation and monitored in the intensive care unit for at least 7 days
  * Glasgow Coma Score ≤10
  * Patients monitored immobile in the intensive care unit
  * Situations where informed consent can be obtained from the patient's legal representative

Exclusion Criteria:

* • Presence of pre-existing joint contracture, ankylosis, or amputation

  * Patients with severe burns, fractures, or surgical reasons preventing joint movement
  * Patients with a history of neuromuscular disease or spasticity
  * Patients who were immobilized for ≥1 week prior to admission to the intensive care unit
  * Hemodynamic instability situations where measurement is unreliable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients admitted to a tertiary-level intensive care unit who are mechanically ventilated, immobilized, and have impaired consciousness. Eligible participants are patients aged 18 years or older who are expected to remain in the ICU for at least seven days and are unable to mobilize independently due to their clinical condition. Patients with pre-existing joint contractures, neuromuscular diseases, spasticity, amputations, or conditions that preclude safe assessment of joint range of motion are excluded. All participants receive routine ICU care and standard physiotherapy according to institutional protocols, and no additional interventions are introduced for research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Joint Contracture During ICU Stay | From ICU admission to ICU discharge or death, whichever occurs first, assessed prospectively for up to 28 days of ICU stay.
  Development of a new joint contracture, defined as a ≥33% reduction in passive range of motion (PROM) compared with normal reference values, measured using a goniometer.

SECONDARY OUTCOMES:
Time to Joint Contracture Development | From ICU admission to the first documented detection of joint contracture, ICU discharge, or death, whichever occurs first, assessed for up to 28 days.
  Time (in days) from ICU admission to the first detection of joint contracture.

CONTACTS AND LOCATIONS:
Locations (1):
- Fethi Sekin City Hospital, Elâzığ, Elaziğ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No